CLINICAL TRIAL: NCT02130739
Title: Incidence of Transient Horner's Syndrome Following Thoracic Epidural Anesthesia for Mastectomy
Brief Title: Horner's SD After Thoracic Epidural Block
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Sun Young Park, MD, Soonchunhyang University Hospital
Other Study IDs: HS-Tepi
Record Dates: First submitted 2014-04-24; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Horner's Syndrome
Keywords: Anesthesia; Epidural; Thoracic Nerves; Horner syndrome
MeSH Terms: conditions — Horner Syndrome | interventions — Mastectomy; Ropivacaine; Propofol; Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- thoracic epidural anesthesia: thoracic epidural anesthesia following continuous thoracic epidural analgesia for mastectomy
  Interventions: Procedure: thoracic epidural anesthesia; Procedure: mastectomy; Drug: Ropivacaine; Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Procedure: thoracic epidural anesthesia — thoracic epidural anesthesia following continuous thoracic epidural analgesia for mastectomy
Procedure: mastectomy — mastectomy with/without breast reconstruction
Drug: Ropivacaine — Thoracic epidural anesthesia performed using 0.375% or 0.5% ropivacaine
Drug: Propofol — Thoracic epidural anesthesia performed followed by sedation consisting of propofol
Drug: Fentanyl — thoracic epidural analgesia continued; supplemented by a continuous epidural infusion of ropivacaine 0.15%, 2 ml/h with fentanyl 8mcg/h.

SUMMARY:
This study prospectively evaluates the incidence of Horner's syndrome after thoracic epidural anesthesia following continuous thoracic epidural analgesia for mastectomy. The incidence was 1.36% and the mechanism of Horner's syndrome was cephalic spread of the local anesthetic.

DETAILED DESCRIPTION:
Transient Horner's syndrome has been recognized rare complication of epidural anesthesia and the incidence is not exactly well-known in thoracic epidural anesthesia. Therefore, this study prospectively evaluates the incidence of Horner's syndrome after thoracic epidural anesthesia following continuous thoracic epidural analgesia for mastectomy.

Six hundred thirty three Patients, who scheduled for mastectomy with/without breast reconstruction, were eligible for this prospective observational study from September 2010 to December 2013. Thoracic epidural anesthesia performed using 0.375% or 0.5% ropivacaine 15mL followed by sedation consisting of propofol without muscle relaxation. After the operation, thoracic epidural analgesia continued; supplemented by a continuous epidural infusion of ropivacaine 0.15%, 2 ml/h with fentanyl 8mcg/h. At 1 hour, 2hour, 1 day, 2 day and 3 day after the operation, postoperative surveillance consisted of the occurrence of symptoms of Horner's syndrome (miosis, ptosis, and hyperemia) were performed by anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who scheduled for mastectomy with/without breast reconstruction

Exclusion Criteria:

* The patients who had more than one abnormal preoperative clotting parameter either clinical signs of potential bleeding disorders suggested by bruising
* Petechiae, or ecchymosis, or anatomic or neurologic abnormalities
* That is, significant scoliosis or kyphosis, radyculopathy or ptosis
* Unsuccessful catheter placement (impossible to insert a catheter at two vertebral levels)
* Unsuccessful epidural anesthesia (not checkable sensory block)
* Dural perforation or intravascular catheterization

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, who scheduled for mastectomy with/without breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Horner's syndrome | 3 day after the operation

SECONDARY OUTCOMES:
Number of Participants with back pain | 3 day after the operation
Number of Participants with radiating symptoms | 3 day after the operation
  segmental pain or paresthesia corresponded to a dermatome of epidural block spinal root
Number of Participants with numbness | 3 day after the operation
Number of Participants with muscular weakness | 3 day after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University Seoul Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park SY, Chun HR, Kim MG, Lee SJ, Kim SH, Ok SY, Cho A. Transient Horner's syndrome following thoracic epidural anesthesia for mastectomy: a prospective observational study. Can J Anaesth. 2015 Mar;62(3):252-7. doi: 10.1007/s12630-014-0284-9. Epub 2015 Jan 6. PMID 25560203